CLINICAL TRIAL: NCT00618605
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled Dose Escalation Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Adenovirus Serotype 26 HIV-1 Vaccine (Ad26.ENVA.01) in Healthy, HIV-1 Uninfected Adults
Brief Title: Safety of and Immune Response to an Adenoviral HIV-1 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ad26.ENVA.01/IPCAVD-001; 10623 (Registry Identifier: DAIDS ES Registry Number); Ad26.ENVA.01
Record Dates: First submitted 2008-02-18; First posted 2008-02-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventative Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 3 injections of Ad26.ENVA.01 HIV-1 vaccine or placebo at 1 x 10^9 virus particles (VP) given at Days 0, 28, and 168
  Interventions: Biological: Ad26.ENVA.01 HIV-1 vaccine
- 2 (Experimental): 3 injections of Ad26.ENVA.01 HIV-1 vaccine or placebo at 1 x 10^10 VP given at Days 0, 28, and 168
  Interventions: Biological: Ad26.ENVA.01 HIV-1 vaccine
- 3 (Experimental): 3 injections of Ad26.ENVA.01 HIV-1 vaccine or placebo at 1 x 10^11 VP given at Days 0, 28, and 168
  Interventions: Biological: Ad26.ENVA.01 HIV-1 vaccine
- 4 (Experimental): 2 injections of Ad26.ENVA.01 HIV-1 vaccine or placebo at a dose to be determined by the safety data from Arms 1, 2 and 3 given at Days 0 and 168
  Interventions: Biological: Ad26.ENVA.01 HIV-1 vaccine

INTERVENTIONS:
Biological: Ad26.ENVA.01 HIV-1 vaccine — Recombinant adenovirus serotype 26 HIV-1 vaccine

SUMMARY:
Successful control of the HIV epidemic will require a safe and effective vaccine to be developed. A successful vaccine will need to stimulate a widespread immune response. The purpose of this study is to determine the safety of and immune response to an adenovirus serotype HIV vaccine in HIV uninfected adults.

DETAILED DESCRIPTION:
HIV infection continues to spread at pandemic levels throughout the world. Control of this pandemic can only be achieved with the development of a safe and effective preventive HIV vaccine. A vaccine that will prevent HIV infection will elicit a strong immune response from both CD4 and CD8 cells. Recombinant adenovirus serotype vectors have been shown to elicit just such a response. The purpose of this study is to determine the safety and immunogenicity of the recombinant adenovirus serotype 26 preventive HIV-1 vaccine.

This study will last 12 months. Participants will be randomly assigned to one of four arms that will receive different doses of the vaccine or placebo administered via intermuscular injection. Participants in Arms 1, 2, and 3 will all receive 3 injections. Each injection will contain the same dose of vaccine. Arm 4 will receive 2 injections of a dose of vaccine that will be determined by the safety data from Arms 1, 2, and 3. Participants will be enrolled sequentially, from lowest to highest dose of vaccine, into Arms 1, 2, and 3. Arms will begin enrollment only following review of safety data from the previous group. After the Day 42 safety data from Arms 1, 2, and 3 have been reviewed, the dose for Arm 4 will be determined, and enrollment into that arm will begin.

There will be 10 study visits in this study, occurring at baseline and after 0.5, 1, 1.5, 2, 6, 6.5, 7, and 12 months. Participants in Arms 1, 2, and 3 will receive injections on Days 0, 28, and 168. Participants in Arm 4 will receive injections on Days 0 and 168. Participants will be asked to record their temperature and other side effects in a symptom log for 7 days after each injection. Risk reduction/pregnancy prevention counseling will occur at visits 1 through 9, and physical exams and assessments of illness or adverse events will occur at all visits. At most visits, blood, urine, and oral swab collection will occur. At some visits, HIV testing and pregnancy testing will occur.

Once a year for 5 years following study entry, participants will attend a study visit or will be contacted by study staff by telephone or e-mail for follow-up safety and health monitoring. Some participants will also undergo a blood collection at these visits.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with normal hematological, hepatic and renal functions
* Demonstrated understanding of study
* Willing to receive HIV test results
* HIV-1 and -2 uninfected
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (anti-HCV) negative antibody or negative HCV PCR if anti-HCV is positive
* Appropriate hemoglobin, white blood cell, lymphocyte, and platelet count values as defined in the study protocol
* Certain laboratory values as defined in the study protocol
* Adequate contraception from at least 21 days prior to study entry through visit 10

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first injection. Participants taking corticosteroid nasal spray or topical corticosteroids are not excluded.
* Blood products within 120 days prior to first injection
* Immunoglobulin within 60 days prior to first injection
* Investigational agents within 30 days prior to first injections
* Live attenuated vaccine within 30 days prior to first injection
* Any vaccine not a live attenuated vaccine within 14 days prior to first injection
* Any clinically significant medical condition that, in the opinion of the investigator, may interfere with the study
* Any medical, psychiatric, occupational, or social condition or responsibility that, in the opinion of the investigator, would interfere with the study
* Serious adverse reaction to vaccines. Participants who had a nonanaphylactic adverse reaction to pertussis vaccine as a child are not excluded.
* Known autoimmune disease
* Known immunodeficiency
* Asthma other than mild and/or well-controlled asthma
* Active syphilis infection. Those fully treated for syphilis over 6 months prior to study entry are not excluded.
* Diabetes mellitus type 1 or 2
* Thyroidectomy or thyroid disease requiring medication within 12 months prior to study entry
* Angioedema in the 3 years prior to study entry if the episodes are considered serious or have required medication within the last 2 years
* Hypertension. More information on this criterion can be found in the protocol.
* Body mass index (BMI) of 40 or higher OR BMI of 35 or greater, if other cardiovascular risk factors. More information on this criterion can be found in the protocol.
* Bleeding disorder
* Malignancy, unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder or occurrence of seizure in the 3 years prior to study entry. Participants who have not required medications or had a seizure for prior 3 years are not excluded.
* Absence of a functional spleen
* Psychiatric condition within the last 3 years. More information on this criterion can be found in the study protocol.
* Individuals at high-risk of acquiring HIV infection
* Presence of pre-existing neutralizing antibodies for Adenovirus 26
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactions to injection | After each injection

SECONDARY OUTCOMES:
Humoral immune responses, such as neutralizing and binding antibodies to HIV and Ad26 | Throughout study
Cell mediated immunity, including T-cell gamma interferon responses and assessment of T-cell responses by flow cytometry | Throughout study
Genotyping | Throughout study
Stored samples may be used to perform additional assays for further evaluation of immunogenicity and to support standardization and validation of new assays such as epitope mapping, flow cytometry, and/or tetramer analysis. | After study follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Study Chair — Brigham and Women's Hospital; Dan Barouch, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center; Raphael Dolin, MD, Study Chair — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hosp. Novel Adenoviral Vector Prophylactic HIV Vaccine Non-Network CRS, Boston, Massachusetts, United States

REFERENCES:
- [Background] Abbink P, Lemckert AA, Ewald BA, Lynch DM, Denholtz M, Smits S, Holterman L, Damen I, Vogels R, Thorner AR, O'Brien KL, Carville A, Mansfield KG, Goudsmit J, Havenga MJ, Barouch DH. Comparative seroprevalence and immunogenicity of six rare serotype recombinant adenovirus vaccine vectors from subgroups B and D. J Virol. 2007 May;81(9):4654-63. doi: 10.1128/JVI.02696-06. Epub 2007 Feb 28. PMID 17329340
- [Background] Liniger M, Zuniga A, Naim HY. Use of viral vectors for the development of vaccines. Expert Rev Vaccines. 2007 Apr;6(2):255-66. doi: 10.1586/14760584.6.2.255. PMID 17408374
- [Background] Roberts DM, Nanda A, Havenga MJ, Abbink P, Lynch DM, Ewald BA, Liu J, Thorner AR, Swanson PE, Gorgone DA, Lifton MA, Lemckert AA, Holterman L, Chen B, Dilraj A, Carville A, Mansfield KG, Goudsmit J, Barouch DH. Hexon-chimaeric adenovirus serotype 5 vectors circumvent pre-existing anti-vector immunity. Nature. 2006 May 11;441(7090):239-43. doi: 10.1038/nature04721. Epub 2006 Apr 16. PMID 16625206
- [Derived] Baden LR, Walsh SR, Seaman MS, Tucker RP, Krause KH, Patel A, Johnson JA, Kleinjan J, Yanosick KE, Perry J, Zablowsky E, Abbink P, Peter L, Iampietro MJ, Cheung A, Pau MG, Weijtens M, Goudsmit J, Swann E, Wolff M, Loblein H, Dolin R, Barouch DH. First-in-human evaluation of the safety and immunogenicity of a recombinant adenovirus serotype 26 HIV-1 Env vaccine (IPCAVD 001). J Infect Dis. 2013 Jan 15;207(2):240-7. doi: 10.1093/infdis/jis670. Epub 2012 Nov 2. PMID 23125444
- [Derived] Barouch DH, Liu J, Peter L, Abbink P, Iampietro MJ, Cheung A, Alter G, Chung A, Dugast AS, Frahm N, McElrath MJ, Wenschuh H, Reimer U, Seaman MS, Pau MG, Weijtens M, Goudsmit J, Walsh SR, Dolin R, Baden LR. Characterization of humoral and cellular immune responses elicited by a recombinant adenovirus serotype 26 HIV-1 Env vaccine in healthy adults (IPCAVD 001). J Infect Dis. 2013 Jan 15;207(2):248-56. doi: 10.1093/infdis/jis671. Epub 2012 Nov 2. PMID 23125443